CLINICAL TRIAL: NCT00933348
Title: A Randomised, Double-blind, Placebo-controlled Study of the Safety and Efficacy of the Fruit-based Product OPAL A for the Treatment of Chronic Venous and Pressure Ulcers.
Brief Title: Safety and Efficacy of the Fruit-based Product OPAL A for the Treatment of Chronic Venous and Pressure Ulcers
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment caused rethink on the study design
Sponsor: Phoenix Eagle Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPAL A-1001
Record Dates: First submitted 2009-07-05; First posted 2009-07-07 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Venous Ulcer; Pressure Ulcer
Keywords: ulcer; venous; pressure; wound; treatment
MeSH Terms: conditions — Varicose Ulcer; Pressure Ulcer; Ulcer; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPAL A plus standard wound care (Active Comparator)
  Interventions: Drug: OPAL A
- Placebo plus standard wound care (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPAL A — OPAL A will be supplied in two formulations: as a Filtrate (0.5 mL per cm2 of ulcer area, applied into the ulcer cavity) and as a Cream (about 1 to 5 g applied as a thin smear on surrounding skin). Both formulations will be applied daily. However, if the ulcer begins to hypergranulate, the OPAL A Filtrate will only be administered once every 72 hours.
  Arms: OPAL A plus standard wound care
Drug: Placebo — Placebo will be supplied in two formulations: as a Filtrate (0.5 mL per cm2 of ulcer area, applied into the ulcer cavity) and as a Cream (about 1 to 5 g applied as a thin smear on surrounding skin). Both formulations will be applied daily. However, if the ulcer begins to hypergranulate, the Placebo Filtrate will only be administered once every 72 hours.
  Arms: Placebo plus standard wound care

SUMMARY:
The purpose of this study is to examine the safety and efficacy of the fruit-based product OPAL A for the treatment of chronic venous and pressure ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Aged ≥ 18 years.
* Presence of either:

  * a venous leg ulcer with a surface area ≥ 2 cm2 and < 25 cm2 (best estimate of debrided wound), OR
  * a Stage II or III pressure ulcer (as per Australian Wound Management Association [AWMA] definitions)
* Able to tolerate compression therapy (for venous ulcer group only)
* Willing and able to provide written informed consent
* Additional inclusion criterion after four-week standard care run-in period:

  * a less than or equal to 25% reduction in wound surface area compared with wound surface area at the screening visit

Exclusion Criteria:

* Another ulcer within 10 cm of the ulcer to be treated
* Patients with diabetes (fasting blood glucose value ≥ 7 mmol/L or random blood glucose > 11 mmol/L) that in the opinion of the investigator is uncontrolled
* Ankle-brachial pressure index of < 0.8 (participants with venous ulcers only)
* Alanine transaminase (ALT) or aspartate transaminase (AST) levels 3X the upper limit of normal
* Any dermatologic condition or disorder (with the exception of dermatitis associated with venous stasis) that may interfere with the appropriate assessment and treatment of the participant's ulcer
* Clinical signs of ulcer infection.
* Current or recent (within the past two weeks) daily treatment with immunosuppressive medications (including oral corticosteroids; inhaled and topical corticosteroids are permitted; topical agents must not be applied within 10 cm of ulcer wound), cytotoxins or anti-inflammatory agents (intermittent non-steroidal anti-inflammatory agent use is permitted)
* Known hypersensitivity to paw paw products
* Pregnancy, planned pregnancy or lactation
* Participation in another clinical trial within one month of study entry
* Another disease or condition that in the opinion of the investigator may jeopardize the safety of the participant or their ability to participate in the study
* Participant previously screened or randomized in this study
* Cognitive impairment that in the opinion of the investigator leaves the participant incapable of providing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | Weekly from Week -4 to Week 12
Physical examination findings and vital signs | Week -6, Day 0 and Weeks 6 and 12
Clinical laboratory assessments (full blood count [FBC], blood chemistry, liver function tests and coagulation parameters) as changed from Day 0 (i.e., baseline/randomization). | Week -6, Day 0, Weeks 3, 6, 12

SECONDARY OUTCOMES:
Time to 50% wound closure | Weekly from Weeks -6 to 12
Time to 100% wound closure | Weekly from Weeks -6 to 12
Proportion of participants with 50% or greater wound closure, or 100% wound closure at 12 weeks | Weekly from Weeks -6 to 12
Percentage change in wound surface area at 12 weeks | Weekly from Weeks -6 to 12
Participant's assessment of pain during wound dressing and wound pain in the 24 hours before each study visit (assessed using the McGill short-form pain survey) | Weekly from Week 0 to 12
Quality of life (QoL) scores and health state (for determination of quality-adjusted life years [QALYs]; assessed using the SF-12 health survey and the McGill short-form pain survey) | Day 0 and Weeks 6 and 12
Participant's and clinician/nurse overall satisfaction with treatment | Weeks 6 and 12
Use of health care resources/informal care | Day 0 and Weekly from Week 1 to 12

CONTACTS AND LOCATIONS:
Overall Officials: Michael Woodward, FRACP, Principal Investigator — Austin Health, Aged Care Services, Medical and Cognitive Research Unit
Locations (1):
- Austin Health, Aged Care Services, Medical and Cognitive Research Unit, Heidelberg West, Victoria, Australia